CLINICAL TRIAL: NCT00172029
Title: Study Comparing Full-dose Radiotherapy Versus Reduced Dose in the Management of Bone Metastasis in Patients With Breast Cancer Receiving Zoledronic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446ETR01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer With Metastatic Bone Disease
Keywords: Zoledronic acid; Radiotherapy; Bone pain; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

ARMS (2):
- ZOL446 Standard radiotherapy dosage (Experimental)
  Interventions: Drug: Zoledronic acid
- ZOL446 Low radiotherapy dosage (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
The aim of this prospective, randomized, open-label, multicentric clinical study is to assess the effícacy and tolerability of zoledronic acid 4 mg IV infused over 15 minutes every 4 weeks for a total of 6 infusions, in combination with standard or reduced dose radiotherapy in patients with breast cancer and metastatic bone disease associated with pain.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years.
* Histologically confirmed diagnosis of breast cancer with at least one bone metastases.
* Radiologically documented solitary or multiple osteolytic or osteoblastic lesions in axial skeleton or in the extremities in which radiotherapy is indicated.
* Pain and/or analgesic score ≥ 3 (see section 3.5.2) at the bone site to be irradiated.
* ECOG performance status ≤ 2.
* Life expectancy more than 6 months.

Exclusion Criteria:

* Patients in whom the target lesion(s) is not detectable by conventional techniques (i.e. X-rays MRI or CT scan).
* Presence of pathological fracture in the target lesion(s).
* Prior irradiation of the painful area(s) to be irradiated.
* Known hypersensitivity to zoledronic acid or other biphosphonates.
* Previous treatment with bisphosphonates for the current disease; any treatment with biphosphonates for other indications should anyway have been discontinued at least two years before randomization into the study.
* Skeleton-related complications (e.g., pathological fractures, orthopedic intervention to treat or stabilize an osteolytic defect, spinal cord compression) during the last 3 weeks prior to the first infusion of trial medication.
* Change in anticancer therapy within the 2 weeks prior to screening assessments and/or test treatment start.
* Patients with severe renal function (serum creatinine > 400 umol/l or > 4.5 mg/dl or calculated creatinine clearance ≤ 30 ml/minute) or with prior renal transplantation. Creatinine clearance will be calculated using the following formula:

Creatinine clearance = (140-age[yr])(body weight [kg]) x 0.85 (72) (serum creatinine [mg/dL]) or Creatinine clearance = (140-age[yr])(body weight [kg]) x 0.85 (0.814) (serum creatinine [µmol/L])

* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L).
* Patients with clinically symptomatic brain metastases
* Bone metabolism disorder, e.g. Paget disease, primary hyperparathyroidism
* Serious intercurrent illness other than breast cancer that can interfere with the evaluation of the effect of the therapy.
* Pregnancy and lactation.
* Women of childbearing potential not on an effective form of contraception.
* Known history or present abuse of alcohol or drugs (accepted social alcohol usage will not exclude the patient)
* Patients who, in the opinion of the investigator, are unlikely to cooperate fully during the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-04; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients showing complete response in bone pain palliation without having any analgesic treatment | day 5, 12, 29; week 8, 12, 16, 20 & 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kayseri
  - Novartis Investigative Site, Trabzon